CLINICAL TRIAL: NCT00236080
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Multiple-Dose Plasma Concentration-Time Profiles of Armodafinil (150, 200, and 250 mg) and PROVIGIL® (200 mg) in Patients With Chronic Shift Work Sleep Disorder
Brief Title: Study of the Efficacy and Multiple-Dose Plasma Concentration-Time Profiles of Armodafinil and PROVIGIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor's Medical Expert, Cephalon
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/3045/CM/US
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Shift Work Sleep Disorder
MeSH Terms: interventions — Modafinil

ARMS (5):
- 1 (Experimental): PROVIGIL 200 mg/day
  Interventions: Drug: PROVIGIL 200 mg
- 2 (Experimental): Armodafinil 250 mg/day
  Interventions: Drug: Armodafinil 250 mg
- 3 (Experimental): Armodafinil 200 mg/day
  Interventions: Drug: Armodafinil 200 mg
- 4 (Experimental): Armodafinil 150 mg/day
  Interventions: Drug: Armodafinil 150 mg
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PROVIGIL 200 mg — PROVIGIL 200 mg/day
  Arms: 1
Drug: Armodafinil 250 mg — Armodafinil 250 mg/day
  Arms: 2
Drug: Armodafinil 200 mg — Armodafinil 200 mg/day
  Arms: 3
Drug: Armodafinil 150 mg — Armodafinil 150 mg/day
  Arms: 4
Drug: Placebo — Matching placebo tablets
  Arms: 5

SUMMARY:
The purpose of the study is to compare the overnight efficacy and plasma concentration-time profiles of armodafinil and PROVIGIL, after multiple doses, in patients with excessive sleepiness associated with chronic Shift Work Sleep Disorder (SWSD).

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Multiple-Dose Plasma Concentration-Time Profiles of Armodafinil and PROVIGIL in Patients with Chronic Shift Work Sleep Disorder

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* The patient speaks and writes in English.
* The patient is a man or woman of any ethnic origin aged 18 through 65 years.
* The patient is in good health as determined by a medical and psychiatric history, medical examination, serum chemistry, and hematology.
* The patient has a diagnosis of SWSD according to the International Classification of Sleep Disorders (ICSD) criteria, and must have had excessive sleepiness during night shifts for at least 3 months.
* The patient must be planning to work at least 3 to 5 nights (per week), of which at least 3 nights will be consecutive.
* The patient must work night shifts that include at least 6 hours between 2200 and 0800 (+30 minutes) and be no longer than 12 hours (+30 minutes) in duration.
* The patient has a mean sleep latency of 6 minutes or less as determined by the MSLT (average of naps at 0100, 0300, 0500, and 0700).
* The patient has a Clinical Global Impression of Severity of Illness (CGI-S) rating of 4 or more as it pertains to sleepiness during night shifts including the commute from work.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include abstinence, barrier method with spermicide, steroidal contraceptive (oral, transdermal, implanted and injected) in conjunction with a barrier method, and intrauterine device (IUD).
* The patient is willing to comply with study restrictions and remain at the clinic overnight as required.
* The patient may have been prescribed PROVIGIL or stimulant therapy for their sleep disorder; however, they must have undergone a washout period of at least 7 days prior to screening assessments done at the second screening visit.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* The patient has any clinically significant medical or psychiatric conditions (treated or untreated).
* The patient has a probable diagnosis of a current sleep disorder other than SWSD.
* The patient consumes caffeine including coffee, tea, and/or other caffeine-containing beverages or foods averaging more than 600 mg of caffeine/day within 2 weeks of the start of study drug administration.
* The patient has medically unexplainable positive urine drug screen (UDS) result at the screening visit.
* The patient has clinically significant deviation from normal in clinical laboratory results, vital signs, or physical examination.
* The patient has received any investigational drug within 30 days or 5 half-lives (whichever is longer) before study drug administration, or in the case of a new chemical entity, 3 months or 5 half-lives (whichever is longer) before study drug adminstration.
* The patient used any prescription drugs disallowed by the protocol or clinical significant use of over-the-counter (OTC) drugs within 7 days before the second screening/baseline visit.
* The patient has any disorder (including gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion.
* The patient has known or suspected hypersensitivity to stimulants and/or modafinil or any ingredient present in the study drug.
* The patient has a history (within the past 5 years) of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual or Mental Disorders of the American Psychiatric Association, Fourth Edition, Text Revision (DSM-IV-TR).
* The patient is a pregnant or lactating woman.
* The patient has donated, within 56 days prior to study drug administration, any blood or plasma in excess of 450 mL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-08; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Neibler, DO, Study Director — Cephalon
Locations (20):
- United States (20):
  - Psypharma Clinical Research, Phoenix, Arizona
  - PsyPharma Clinical Tucson, Tucson, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Pacific Sleep Medicine Service, Los Angeles, California
  - Pacific Sleep Medicine Service, San Diego, California
  - BMR HealthQuest, San Diego, California
  - Stanford University, Stanford, California
  - Neurotrials Research, Atlanta, Georgia
  - SLEEPMED, Inc., Macon, Georgia
  - Henry Lahmeyer, MD, Northfield, Illinois
  - Vince and Associates Clinical, Overland Park, Kansas
  - Center for Sleep/Wake Disorder, Chevy Chase, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Rsch Center of Nevada, Las Vegas, Nevada
  - Clinilabs / Sleep Disorders In, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - St. Vincent Mercy Medical Cent, Toledo, Ohio
  - Consolidated Clinical Trials, Pittsburgh, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Radiant Research Salt Lake, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 centers in the US. First participant enrolled: 7 September 2005/ Last participant last visit: 1 December 2005
Pre-assignment Details: 2 male participants withdrew after randomization but prior to receiving study drug (1 for noncompliance and 1 at the request of the sponsor)
Groups:
- PROVIGIL 200 mg/Day: PROVIGIL 200 mg once daily only on nights worked
- Armodafinil 250 mg/Day: Armodafinil 250 mg once daily only on nights worked
- Armodafinil 200 mg/Day: Armodafinil 200 mg once daily only on nights worked
- Armodafinil 150 mg/Day: Armodafinil 150 mg once daily only on nights worked
- Placebo: Matching placebo tablets once daily only on nights worked
Period: Overall Study
Arm/Group | PROVIGIL 200 mg/Day | Armodafinil 250 mg/Day | Armodafinil 200 mg/Day | Armodafinil 150 mg/Day | Placebo
Started | 29 | 28 | 27 | 25 | 27
Completed | 27 | 27 | 22 | 23 | 26
Not Completed | 2 | 1 | 5 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROVIGIL 200 mg/Day | Armodafinil 250 mg/Day | Armodafinil 200 mg/Day | Armodafinil 150 mg/Day | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 27 | 25 | 27 | 136
Age Categorical [Number; unit: participants] — 2 male participants withdrew after randomization but prior to receiving study drug (1 for noncompliance and 1 at the request of the sponsor)
  participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 29 | 28 | 26 | 25 | 26 | 134
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (8.92) | 34.3 (9.87) | 34.5 (7.60) | 38.3 (12.83) | 38.0 (9.83) | 36.3 (9.90)
Gender [Number; unit: participants] — 2 male participants withdrew after randomization but prior to receiving study drug (1 for noncompliance and 1 at the request of the sponsor)
  participants
    Female | 18 | 12 | 13 | 8 | 6 | 57
    Male | 11 | 16 | 13 | 17 | 20 | 77
Region of Enrollment [Number; unit: participants] — 2 male participants withdrew after randomization but prior to receiving study drug (1 for noncompliance and 1 at the request of the sponsor)
  participants
    United States | 29 | 28 | 26 | 25 | 26 | 134

OUTCOME MEASURES:

1. Primary Outcome: Multiple Sleep Latency Test (MSLT)
Description: The Multiple Sleep Latency Test (MSLT) is an objective assessment of sleepiness that measures the likelihood of falling asleep. Five 20-minute (maximum) MSLT naps were performed (at 2300, 0100, 0300, 0500, and 0700) at both the screening/baseline assessment visit (Visit 2) and at endpoint (Visit 4). Each nap was terminated after 20 minutes if no sleep occurred. Sleep latency was measured as the elapsed time from lights out to the first epoch scored as sleep.
Time Frame: Endpoint (Visit 4) change from baseline (Visit 2)
Population: * 1 Placebo Patient did not have an MSLT but did complete the other Primary Measure (PVT) and other requirements. This patient was termed a "Completer".
  * 1 Patient in the "Armodafinil 200 mg/day group" had an MSLT performed but then discontinued the study drug before reaching the study endpoint and was termed a "Non-Completer" for the Study.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | PROVIGIL 200 mg/Day | Armodafinil 250 mg/Day | Armodafinil 200 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 27 | 27 | 23 | 23 | 25
Minutes | 2.0 (3.05) | 3.7 (4.33) | 3.7 (5.07) | 2.7 (4.24) | 1.1 (3.76)
Statistical Analysis 1: Comparison: PROVIGIL 200 mg/Day vs Armodafinil 250 mg/Day vs Armodafinil 200 mg/Day vs Armodafinil 150 mg/Day vs Placebo; Sample size requirements were not based on statistical considerations. The null hypothesis was Ho: μplacebo = μ150 = μ200 = μ250 = μprovigil versus Ha: at least 2 of the means are different, where μ represented the change from baseline to the endpoint; Test type: Non-Inferiority or Equivalence — Number of participants analyzed was determined by those participants who had at least 1 postbaseline efficacy assessment. Sample size requirements were not based on statistical considerations. There were 20 patients in each of the 5 treatment groups, for a total of 100 patients. It is expected that the sample size will provide sufficient information for describing the specified evaluations; p = 0.1236, ANCOVA — The p-value of Overall Treatment to Placebo; This analysis adjusted for the difference among the treatment groups at baseline

2. Primary Outcome: Psychomotor Vigilance Task (PVT)
Description: The computer-based PVT took 10 minutes to complete and measured reaction time stimulus in milliseconds. The reaction time consisted of the digits 000 initially appearing in a window on the PVT device, after which the 3-digit numbers increased in milliseconds until the response button was pressed by the patient. The resulting number at the button press was the reaction time in milliseconds. There was a variable 1- to 10-second interstimulus interval. After pressing the button in response to each stimulus, the button was released and the patient awaited the next stimulus.
Time Frame: Endpoint (Visit 4) change from baseline (Visit 2)
Population: Of the patients who completed the study, 1 patient in the PROVIGIL 200 mg/day treatment group and 1 patient in the Armodafinil 150 mg/day treatment group did not complete their PVT assessment.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | PROVIGIL 200 mg/Day | Armodafinil 250 mg/Day | Armodafinil 200 mg/Day | Armodafinil 150 mg/Day | Placebo
Number analyzed (Participants) | 26 | 27 | 22 | 22 | 26
Milliseconds | -16.5 (27.58) | -29.8 (38.35) | -37.4 (63.16) | -33.1 (44.52) | 2.4 (34.52)
Statistical Analysis 1: Comparison: PROVIGIL 200 mg/Day vs Armodafinil 250 mg/Day vs Armodafinil 200 mg/Day vs Armodafinil 150 mg/Day vs Placebo; Sample size requirements were not based on statistical considerations. The null hypothesis was Ho: μplacebo = μ150 = μ200 = μ250 = μprovigil versus Ha: at least 2 of the means are different, where μ represented the change from baseline to the endpoint; Test type: Non-Inferiority or Equivalence — Using the adjusted p value from Tukey's least significant difference (LSD) test for armodafinil at 200 mg/day. Sample size requirements were not based on statistical considerations. There were 20 patients in each of the 5 treatment groups, for a total of 100 patients; p = 0.0945, ANCOVA — The p-value of Overall Treatment to Placebo

ADVERSE EVENTS:
Arm/Group | PROVIGIL 200 mg/Day | Armodafinil 250 mg/Day | Armodafinil 200 mg/Day | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/26 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 5/29 | 8/28 | 9/26 | 4/25 | 3/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PROVIGIL 200 mg/Day (N=29) | Armodafinil 250 mg/Day (N=28) | Armodafinil 200 mg/Day (N=26) | Armodafinil 150 mg/Day (N=25) | Placebo (N=26)
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 4 | 3 | 3 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
In analyzing the PVT data, it was discovered that data transfer errors had occurred at certain study centers. The ability to interpret the efficacy results from this study is limited, and the findings should be considered inconclusive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days